CLINICAL TRIAL: NCT02529774
Title: Efficacy and Safety of Alternating Systemic and Hepatic Artery Infusion Therapy Versus Systemic Chemotherapy Alone As Adjuvant Treatment After Resection of Liver Metastases From Colorectal Cancer: A Randomized, Parallel-Group, Open-Labelled, Active-Controlled Phase II/III Trial in China
Brief Title: Alternating Systemic and Hepatic Artery Infusion Therapy As Adjuvant Treatment After Resection of Liver Metastases From Colorectal Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ye Xu (Other)
Responsible Party: Sponsor-Investigator, Ye Xu, Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1507149-6
Record Dates: First submitted 2015-08-18; First posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Resected Liver Metastases From Colorectal Cancer
MeSH Terms: interventions — Floxuridine; Heparin; Oxaliplatin; Capecitabine; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Systemic Chemotherapy plus Hepatic Artery Infusion (HAI) (Experimental)
  Interventions: Drug: Floxuridine (FUDR),Dexamethasone (DXM), Heparin in combination with Oxaliplatin and Capecitabine (CapeOX) or in combination with Oxaliplatin and Leucovorin and 5-FU (mFOLFOX6)
- Systemic Chemotherapy (Active Comparator)
  Interventions: Drug: Oxaliplatin and Capecitabine (CapeOX) or Oxaliplatin and Leucovorin and 5-FU (mFOLFOX6)

INTERVENTIONS:
Drug: Floxuridine (FUDR),Dexamethasone (DXM), Heparin in combination with Oxaliplatin and Capecitabine (CapeOX) or in combination with Oxaliplatin and Leucovorin and 5-FU (mFOLFOX6) — Hepatic Artery Infusion for four cycles:
  Floxuridine (FUDR) 500mg/d, Day 1-2; DXM 1mg/day added to FUDR 2-day infusion; Heparin 1000U/day added to FUDR 2-day infusion
  In combination with Systemic Chemotherapy CapeOX for 8 cycles:
  Oxaliplatin 130 mg/m^2 iv over 2 hours, Day 1. Capecitabine 850mg/m^2/d PO Bid, given in the morning and evening, Day 1-14
  Or in combination with Systemic Chemotherapy mFOLFOX6 for 12 cycles:
  Oxaliplatin 85mg/m^2 IV over 2 hours, Day 1. Leucovorin 400mg/m^2 IV over 2 hours, Day 1 5-fluorouracil (FU) 400mg/m^2 IV and then 2400mg/m^2 over 48 hours IV continuous infusion. Day 1
  Arms: Systemic Chemotherapy plus Hepatic Artery Infusion (HAI)
Drug: Oxaliplatin and Capecitabine (CapeOX) or Oxaliplatin and Leucovorin and 5-FU (mFOLFOX6) — Systemic Chemotherapy CapeOX alone for 8 cycles:
  Oxaliplatin 130 mg/m^2 iv over 2 hours, Day 1. Capecitabine 850mg/m^2/d PO Bid, given in the morning and evening, Day 1-14
  Or Systemic Chemotherapy mFOLFOX6 alone for 12 cycles:
  Oxaliplatin 85mg/m^2 IV over 2 hours, Day 1. Leucovorin 400mg/m^2 IV over 2 hours, Day 1 5-fluorouracil (FU) 400mg/m^2 IV and then 2400mg/m^2 over 48 hours IV continuous infusion. Day 1
  Arms: Systemic Chemotherapy

SUMMARY:
This adaptive seamless Phase II/III trial is to compare the efficacy and safety of adjuvant systemic chemotherapy (SCT) with or without hepatic arterial infusion (HAI) after complete hepatic resection for Chinese patients with metastatic colorectal cancer.

ELIGIBILITY:
Diagnosis Criteria:

All patients should have histologically confirmed colorectal adenocarcinoma with hepatic metastases and primary tumours completely resected during the operation and with colorectal metastatic to the liver confirmed pathologically after the operation as well as with negative surgical margin.

Main criteria for inclusion:

* Aged 18-75 years
* Diagnosed as colorectal adenocarcinoma which only spread to the liver and with no extra-hepatic metastases
* Prior curative resection of primary tumours (R0 resection) or concurrent feasible curative resection of primary tumours and hepatic metastases (R0 resection is met)
* Performance status ECOG 0-1
* No serious complication occurred during or after metastases resection and affected subsequent treatment.
* Hematology: White blood count ≧ 4.0X10^9/L, Absolute neutrophil count ≧1.5X10^9/L, Platelet count ≧ 100 X10^9/L, Hemoglobin ≧ 100g/L
* Blood biochemistry: Total bilirubin ≦2mg/dL , Direct bilirubin equal or less than 1.5 times upper limit of normal (ULN), Alanine aminotransferase (ALT) no greater than 2.5 times ULN, Aspartate aminotransferase (AST) no greater than 2.5 times ULN, Serum creatinine no greater than ULN, or glomerular filtration rate equal or greater than 60 mL/min/1.73m^2
* Not pregnant or nursing at present
* Fertile patients must use effective contraception
* Able to withstand major operative procedure
* No prior or concurrent malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of any organ
* No prior hepatic artery infusion therapy with 5-FU or floxuridine
* No prior systemic chemotherapy for metastatic disease
* No other concurrent chemotherapy
* Able to understand and sign off informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2015-09; Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 5-year
  Overall survival will be measured from the date of randomization up to the date of death of any cause
Liver Relapse-Free Survival Rate | 3-year
  Liver Relapse-Free Survival (LRFS) is defined as the interval from the date of randomization to the date of liver localized metastatic relapse (with the exception of curatively treated non-melanoma skin cancer or carcinoma in situ of the cervix) or death from any cause whichever occurs first.

SECONDARY OUTCOMES:
Disease free survival | 3-year
  DFS is defined as the time interval from the date of randomization to the time of the first relapse at any site, death from any cause, or last recorded follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Xu, Dr., Principal Investigator — Fudan University Shanghai Cancer Center China
Locations (1):
- Fudan University Shanghai Cancer Center China, Shanghai, Shanghai Municipality, China